CLINICAL TRIAL: NCT02385292
Title: Randomized, Controlled, Crossover, Multicenter Trial Comparing Quality of Tears Produced by Nasal Neurostimulation Versus Sham for Dry Eye
Brief Title: Multicenter Trial Evaluating Quality of Tears Produced by Nasal Neurostimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oculeve, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: OCUN-003
Record Dates: First submitted 2015-03-02; First posted 2015-03-11 (Estimated); Results first posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intranasal then Extranasal Application (Experimental): Intranasal application of the Oculeve Intranasal Lacrimal Neurostimulator followed by extranasal application of the Oculeve Intranasal Lacrimal Neurostimulator.
  Interventions: Device: Oculeve Intranasal Lacrimal Neurostimulator
- Extranasal then Intranasal Application (Active Comparator): Extranasal application of the Oculeve Intranasal Lacrimal Neurostimulator followed by Intranasal application of the Oculeve Intranasal Lacrimal Neurostimulator.
  Interventions: Device: Oculeve Intranasal Lacrimal Neurostimulator

INTERVENTIONS:
Device: Oculeve Intranasal Lacrimal Neurostimulator — The Oculeve Intranasal Lacrimal Neurostimulator applies a small electrical current to gently activate the body's natural tear production system.

SUMMARY:
The objectives of this study are:

* To compare the change in levels of tear proteins and inflammatory mediators pre and post administration between the intranasal and extranasal applications
* To compare the goblet cell count following application between the intranasal and extranasal applications
* To compare fluorescein tear clearance with the application of the device intranasally and extranasally applications

DETAILED DESCRIPTION:
In this study, subjects will participate for three study days during up to a 44 day period, consisting of a screening examination to determine eligibility on one day and study applications on two different days. There are two applications, intranasal and extranasal. Subjects will receive both applications, in random sequence, one at each of the two application days (Visit 2 and Visit 3). The two applications consist of:

* Active intranasal device application
* Active extranasal device application

ELIGIBILITY:
Inclusion Criteria:

* Bilateral dry eyes
* Capable of providing written informed consent

Exclusion Criteria:

* Chronic or recurring epistaxis (nosebleeds)
* Blood coagulation disorder
* Uncontrolled or poorly controlled diabetes
* Heart or pulmonary disease
* Females who are pregnant, planning a pregnancy or nursing

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-05-31 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lewis, MD, Principal Investigator — Grutzmacher, Lewis & Sierra
Locations (2):
- United States (2):
  - Grutzmacher, Lewis & Sierra, Sacramento, California
  - Baylor College of Medicine, Department of Ophthalmology, Houston, Texas

REFERENCES:
- [Derived] Gumus K, Schuetzle KL, Pflugfelder SC. Randomized Controlled Crossover Trial Comparing the Impact of Sham or Intranasal Tear Neurostimulation on Conjunctival Goblet Cell Degranulation. Am J Ophthalmol. 2017 May;177:159-168. doi: 10.1016/j.ajo.2017.03.002. Epub 2017 Mar 14. PMID 28302532

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During transfer and acquisition of study record by sponsors, no study data has been located and all efforts to locate study data have been exhausted. Therefore, no study data is available to report at this time.
Period: Overall Study
Arm/Group | Intranasal Then Extranasal Application | Extranasal Then Intranasal Application
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: During transfer and acquisition of study record by sponsors, no study data has been located and all efforts to locate study data have been exhausted. Therefore, no study data is available to report at this time.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Then Extranasal Application | Extranasal Then Intranasal Application | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous [unit: years]
Sex: Female, Male [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Fluorescein Tear Clearance With Application
Time Frame: Day 1
Population: as for baseline characteristics
Groups:
- Intranasal Application: Intranasal application of the Oculeve Intranasal Lacrimal Neurostimulator.
- Extranasal Application: Extranasal application of the Oculeve Intranasal Lacrimal Neurostimulator.
Arm/Group | Intranasal Application | Extranasal Application
Number analyzed (Participants) | 0 | 0

2. Other Pre Specified Outcome: Level of Tear Proteins Pre and Post Administration
Time Frame: Day 1
Population: as for baseline characteristics
Arm/Group | Intranasal Application | Extranasal Application
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Level of Inflammatory Mediators Pre and Post Administration
Time Frame: Day 1
Population: as for baseline characteristics
Arm/Group | Intranasal Application | Extranasal Application
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Goblet Cell Count Following Application
Time Frame: Day 1
Population: as for baseline characteristics
Arm/Group | Intranasal Application | Extranasal Application
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: During transfer and acquisition of study record by sponsors, no study data has been located and all efforts to locate study data have been exhausted. Therefore, no study data is available to report at this time.
Arm/Group | Intranasal Application | Extranasal Application
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
During transfer and acquisition of study record by sponsors, no study data has been located and all efforts to locate study data have been exhausted. Therefore, no study data is available to report at this time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator or other study-related personnel may not disclose to anyone or use any data, information, or materials related to this clinical trial without the express written consent of Oculeve.